CLINICAL TRIAL: NCT06529302
Title: Association of Axillary Lymph Node Dissection With Oncological Outcomes in Patients With Residual Micrometastases After Neoadjuvant Chemotherapy: The OPBC-07/microNAC Study
Brief Title: The OPBC-07/microNAC Study
Status: Active, not recruiting | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-00186; bb24Weber
Record Dates: First submitted 2024-07-25; First posted 2024-07-31 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Breast Cancer
Keywords: Neoadjuvant chemotherapy; Axillary lymph node dissection; Residual micrometastases
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this multicenter retrospective cohort study is to determine the safety of omission of axillary lymph node dissection in patients with residual micrometastases after neoadjuvant chemotherapy.

DETAILED DESCRIPTION:
Chemotherapy before surgery, known as neoadjuvant chemotherapy (NAC), is often used to treat patients with advanced breast cancer or aggressive early-stage breast cancer. Research shows that about one in four early-stage breast cancer patients receives this treatment.

For patients undergoing NAC, standard of care includes checking the lymph nodes under the arm (axillary lymph nodes) using a procedure called Sentinel lymph node biopsy to determine if the cancer has spread. In cases where the cancer has spread to the lymph nodes but then shrinks or disappears after chemotherapy, special techniques like dual tracer mapping, targeted axillary dissection, or the Marking Axillary Lymph Nodes with Iodine Seeds procedure are used to ensure accurate biopsy results.

For patients whose cancer shrinks completely in the lymph nodes, it is generally safe to skip further surgery to remove more lymph nodes, a procedure called axillary lymph node dissection (ALND). However, if cancer remains in the lymph nodes, more lymph nodes are typically removed because there is a high chance that cancer is still present.

An increasing number of surgeons are starting to omit ALND, especially when only tiny amounts of cancer (micrometastases) remain. To ensure this practice is safe, real-world data on patient outcomes over time is needed.

This multicenter retrospective cohort study aims to assess the safety of omitting ALND in patients with residual micrometastases after NAC for breast cancer. The study analyzes data of breast cancer patients treated between 2013 and 2024 at more than 50 centers that are part of the Oncoplastic Breast Consortium.

The results of this study will provide valuable information to help doctors determine the best treatment approach for their patients.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive women and men aged 18 years or older with a diagnosis of stage I-III breast cancer (any histological and receptor subtype)
* For Clinically Node negative (cN0) at presentation: any axillary staging technique including palpation is allowed. Dual tracer mapping is not required for Sentinel Lymph Node Biopsy (SLNB)
* For Clinically Node positive (cN+) at presentation: Biopsy proven confirmation is required. Staging techniques include: SLNB with dual mapping or targeted axillary dissection (Targeted Axillary Dissection, TAD: imaging-guided localization of sampled node in combination with Sentinel Lymph Node procedure with or without dual mapping) or the Marking Axillary Lymph Nodes with Iodine Seeds (MARI) procedure
* Completed neoadjuvant chemotherapy
* Residual micrometastases detected on SLNB or TAD or MARI (on frozen section or final pathology)
* Concomitant presence of Isolated Tumor Cells (ITCs) and micrometastases in other sentinel lymph nodes is allowed
* Received axillary treatment with completion axillary lymph node dissection (ALND), axillary Radiotherapy (ART), both or none
* At least 1-year follow-up (inclusion should end in May 2023)
* Had surgery at any time point until May 2023 at the latest
* Prior history of stage I-III (not stage IV) breast cancer is allowed

Exclusion Criteria:

* Did not undergo SLNB/TAD/MARI (e.g., went straight to ALND or ART)
* Presence of ITCs alone or macrometastases on the sentinel nodes (or TAD nodes or MARI node)
* Stage IV disease at presentation
* Inflammatory breast cancer at presentation
* Neoadjuvant endocrine therapy
* Micrometastases detected by One-step nucleic acid amplification (OSNA)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study assesses consecutive patients with residual micrometastases after neoadjuvant chemotherapy, treated with or without axillary dissection. The data originate from participating Oncoplastic Breast Consortium (OPBC) centers as well as from the US and Brazil, and have been collect within the clinical routine between 2013 and 2024.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2024-05-15 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
5-year rate of any axillary recurrence | 5 years
  Assessment of the incidence of any axillary recurrence, which is defined as isolated or combined with local or distant recurrence.
5-year rate of isolated axillary recurrence | 5 years
  Assessment of the incidence of isolated axillary recurrence.
Comparison of 5-year rate of axillary recurrence in patients treated with and without axillary dissection | 5 years
  The incidence of axillary recurrence is compared between patients that were treated with and without axillary dissection.

SECONDARY OUTCOMES:
Proportion of patients with additional micro- and macrometastases removed by axillary lymph node dissection | 5 years
  Assessment of the proportion of patients with additional micro- and macrometastases that were removed by axillary lymph node dissection.
5-year rates of locoregional and any invasive recurrence | 5 years
  Assessment of the incidence of locoregional and any invasive recurrence.
Comparison of 5-year rate of locoregional and any invasive recurrence in patients treated with and without axillary lymph node dissection | 5 years
  The incidence of locoregional and any invasive recurrence is compared between patients that were treated with and without axillary lymph node dissection.

CONTACTS AND LOCATIONS:
Overall Officials: Walter Paul Weber, Prof. Dr., Principal Investigator — University Hospital, Basel, Switzerland
Locations (84):
- United States (19):
  - Valleywise Health Medical Center, Phoenix, Arizona
  - Cedars-Sinai Medical Center, Los Angeles, California
  - University of California, San Francisco, California
  - Providence Saint John's Cancer Institute, Santa Monica, California
  - University of Miami, Coral Gables, Florida
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - NYU Langone Health, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Montefiore Medical Center, New York, New York
  - University of Rochester, Rochester, New York
  - Duke University, Durham, North Carolina
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - MD Anderson Cancer Center, Houston, Texas
  - Swedish Cancer Institute, Seattle, Washington
  - University of Washington, Seattle, Washington
- Sanatorio Modelo Quilmes, Quilmes, Argentina
- Chris O'Brien Lifehouse (COBL), Sydney, Australia
- Austria (2):
  - Ordensklinikum Linz GmbH, Linz
  - Medical University of Vienna Chirurgie, Vienna
- Brazil (9):
  - Hospital de Base do Distrito Federal, Brasília
  - Sirio Libanes Hospital Brasilia, Brasília
  - Hospital Nossa Senhora das Graças, Curitiba
  - Hospital Geral de Fortaleza, Fortaleza
  - Instituto do Cancer do Ceará, Fortaleza
  - Instituto de Mastologia e Oncologia, Goiânia
  - Hospital de Câncer Araújo Jorge, Goiânia
  - Sirio Libanes Hospital, São Paulo
  - Instituto D'OR de Pesquisa e Ensino, São Paulo
- Sir Mortimer B. Davis Jewish General Hospital, Montreal, Canada
- Chile (2):
  - Arturo Lopez Perez Foundation, Providencia
  - Institute of Radiation Medicine, Vitacura
- Clinical Hospital Center Rijeka, Rijeka, Croatia
- Mansoura oncology center, Al Mansurah, Egypt
- Germany (5):
  - University Hospital Augsburg, Augsburg
  - University Hospital Düsseldorf, Düsseldorf
  - KEM | Clinics Essen-Mitte, Essen
  - University Hospital Heidelberg, Heidelberg
  - University Hospital Lübeck, Lübeck
- Greece (2):
  - University General Hospital of Heraklion, Heraklion
  - Athens Medical Center, Marousi
- Sheba Medical Center, Ramat Gan, Israel
- Italy (5):
  - Insituto Europeo di Oncologia, Milan
  - University Hospital Federico II, Napoli
  - IOV Padua, Padua
  - Clinici Scientifici Maugeri IRCCS, Pavia
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Roma
- Pauls Stradiņš Clinical University Hospital, Riga, Latvia
- National Cancer Institute, Vilnius, Lithuania
- The Netherlands Cancer Institute - Antoni van Leeuwenhoek Hospital, Amsterdam, Netherlands
- Oslo University Hospital, Oslo, Norway
- Dow University of Health Sciences, Karachi, Pakistan
- Peru (2):
  - Hospital Nacional Guillermo Almenara Irigoyen, La Victoria
  - Instituto Nacional de Enfermedades Neoplasicas, Surquillo
- University Hospital Zielona Gora, Zielona Góra, Poland
- Champalimaud Foundation, Lisbon, Portugal
- N.N. Petrov National Medical Research Center of Oncology, Saint Petersburg, Russia
- AGEL Mammacentrum sv. Agáty, Banská Bystrica, Slovakia
- Institute of Oncology Ljubljana, Ljubljana, Slovenia
- South Korea (4):
  - ASAN Medical Center, Seoul
  - Gangnam Severance Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul
- Spain (3):
  - Hospital del Mar d'Investigacions Mèdiques, Barcelona
  - Clinica Universidad de Navarra, Madrid
  - Hospital Universitario La Paz, ía Mamaria, Madrid
- Capio Saint Göran's Hospital, Stockholm, Sweden
- Switzerland (9):
  - Cantonal Hospital Baden, Baden
  - University Hospital Basel, Basel
  - Campus SLB Sonnenhof AG, Bern
  - Cantonal Hospital Luzern, Lucerne
  - EOC Centro di Senologia della Svizzera Italiana, Lugano
  - Tumor und Brustzentrum Ostschweiz, Sankt Gallen
  - Cantonal Hospital Winterthur, Winterthur
  - Zürich Breast Center, Zurich
  - University Hospital Zürich, Zurich
- Turkey (Türkiye) (4):
  - Gülhane Training and Research Hospital, Ankara
  - Istanbul University Faculty of Medicine, Fatih
  - Marmara University, Istanbul
  - Zonguldak Bülent Ecevit University, Zonguldak
- Cambridge University Hospitals, Cambridge, United Kingdom

REFERENCES:
- [Derived] Montagna G, Alvarado M, Myers S, Mrdutt MM, Sun SX, Sevilimedu V, Barrio AV, van den Bruele AB, Boughey JC, Boyle MK, Crown A, Kesmodel SB, King TA, Kuerer HM, Leisha EC, Moo TA, Weiss A, Williams AD, Parmar P, Diskin B, Hlavin C, Diego EJ, Polidorio N, Abdelwahab K, Banys-Paluchowski M, Kurzeder C, Heidinger M, Goldschmidt M, Schulz A, Heil J, Karadeniz Cakmak G, Pislar N, Riis M, Prakash I, Ovalle V, Ugurlu MU, Franceschini G, Sergeevich EA, Morales J, Lee HB, Galimberti V, Ahn SG, Ryu JM, Muslumanoglu M, Cabioglu N, Yoo TR, Vrancken Peeters MJ, Ferrucci M, Morrow M, Weber WP; microNAC Study Group. Oncological outcomes with and without axillary lymph node dissection in patients with residual micrometastases after neoadjuvant chemotherapy (OPBC-07/microNAC): an international, retrospective cohort study. Lancet Oncol. 2026 Jan;27(1):57-67. doi: 10.1016/S1470-2045(25)00598-4. PMID 41449148